CLINICAL TRIAL: NCT03241407
Title: Effect of a Triclosan-containing Toothpaste as a Preventive Strategy of Peri-implant Experimental Mucositis in Cigarette Smokers: Clinical and Osteo-immunoinflammatory Response in a Randomized Crossover Study.
Brief Title: Triclosan Toothpaste as a Preventive Strategy of Mucositis in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Fernanda Vieira Ribeiro, Professor, Paulista University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Triclosan Mucositis Smoking
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Dental Implants; Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Triclosan

STUDY DESIGN:
Intervention Model Description: This investigation was designed as double-blind, randomized, crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo toothpaste (Placebo Comparator): Fluoride toothpaste will be used by filling the individual silicone stent allowing it to come into contact with the implant area for 2 min.During an experimental 3-week period of undisturbed mechanical plaque accumulation in the implants, implants randomly assigned to Placebo group will be submitted to a chemical plaque control (three times per day) using a Triclosan toothpaste.
  Interventions: Other: Placebo toothpaste
- triclosan/copolymer/fluoride toothpaste (Experimental): triclosan/copolymer/fluoride toothpaste will be used by filling the individual silicone stent allowing it to come into contact with the implant area for 2 min. During an experimental 3-week period of undisturbed mechanical plaque accumulation in the implants, implants randomly assigned to triclosan/copolymer/fluoride group will be submitted to a chemical plaque control (three times per day) using a triclosan/copolymer/fluoride toothpaste.
  Interventions: Other: triclosan/copolymer/fluoride toothpaste

INTERVENTIONS:
Other: Placebo toothpaste — During an experimental 3-week period of undisturbed mechanical plaque accumulation in the implants, implants randomly assigned to Placebo group will be submitted to a chemical plaque control (three times per day) using a placebo toothpaste.
  Arms: Placebo toothpaste
Other: triclosan/copolymer/fluoride toothpaste — During an experimental 3-week period of undisturbed mechanical plaque accumulation in the implants, implants randomly assigned to triclosan/copolymer/fluoride group will be submitted to a chemical plaque control (three times per day) using a triclosan/copolymer/fluoride toothpaste.
  Arms: triclosan/copolymer/fluoride toothpaste

SUMMARY:
The purpose of this trial was to determine the effect of a triclosan-containing toothpaste in the clinical parameters and in the profile of osteo-immunoinflammatory mediators in the peri-implant crevicular fluid (PICF) as a preventive therapy of peri-implant experimental mucositis in cigarette smokers

DETAILED DESCRIPTION:
This study was designed as double-blind, randomized, crossover study to evaluate the influence of a triclosan-containing toothpaste in the profile of osteo-immunoinflammatory mediators in the PICF of smoker individuals and in the clinical measurements during the progression of experimental peri-implant mucositis. This investigation was approved by the ethics committee of Paulista University . Patient recruitment started in July 2013 and was completed by the end of September 2014. Clinical procedures and evaluations were carried out between September 2013 and November 2014. Data entry and statistical analyses were performed in April 2015. All the patients in the study were recruited from the patients referred to Paulista University. Patients were thoroughly informed of the nature, potential risks and benefits of their participation in the study, and they each signed an informed consent document. During this 3-week period, participants were randomly assigned to two groups by a computer-generated list: Triclosan (n=13): triclosan/copolymer/fluoride toothpaste or Placebo (n=13): fluoride toothpaste, by filling the individual silicone stent with the respective toothpaste, according to the experimental group, and allowing it to come into contact with the implant area for 2 min, three times per day. Conventional tooth brushing was performed in the non-stent areas.

After 3 weeks, a professional prophylaxis was performed and a wash-out period of 30 days was established. All patients restarted their optimal mechanical plaque control practices to reach pre-experimental levels of oral cleanliness and gingival/mucosal health. Then, a second experimental 3-week period of undisturbed plaque accumulation around the implants was established and the experimental groups were exchanged. After that, a new professional prophylaxis was performed. Patients were blinded to the therapies.All evaluations (clinical and immunoenzimatic) were performed at baseline, 3, 7, 14 and 21 days of each period of experimental mucositis induction. Levels of osteo-immunoinflammatory mediators were considered primary outcome variable. The number of patients included was based on previous crossover investigations that found differences in the crevicular fluid levels of osteo-immunoinflammatory markers in different clinical status. The same examiner (SPP), who was blinded to the groups, performed all clinical measurements. To perform the intra-examiner calibration, 15 non-study individuals presenting dental implants were selected. The examiner measured the PD of all individuals twice within 24 hours. The intra-class correlation was calculated as 95% reproducibility.

Individual stents were prepared to standardize the location of periodontal probe in order to evaluate the following parameters at four sites of the experimental dental implants at baseline, 3, 7, 14, 21 days follow-ups: 1) plaque index (PI/%): dichotomous plaque index along the mucosal margin around implants, 2) Bleeding on probing (BOP,%):dichotomous index of bleeding during probing around implants, 3) Position of the peri-implant margin (PPM/mm): distance from the stent to the peri-implant margin; 4) Relative clinical attachment level (RCAL/mm): distance from the stent to the bottom of the peri-implant pocket; and 5) Peri-implant Probing depth (PD,mm): calculated by deducting PPM from RCAL.

Levels of interferon, interleukin (IL)-17, IL-1β, IL-10, IL-6, IL-8, tumor necrosis factor (TNF)-α , osteoprotegerin (OPG), osteocalcin (OC), osteopontin (OPN) , matrix metalloproteinase (MMP)-2, MMP-9 , transforming growth factor (TGF)-β , soluble receptor activator of nuclear factor ligand (RANKL) and crosslinked telopeptide of type I collagen (ICTP) in the PICF were determined using the MAGpix™ instrument and Xponent® software . The mean concentration of each mediator was calculated using the individual as a statistical unit and expressed as pg/ml.

All analyses were completed using SAS program release 9.1 . Data were examined for normality using the Kolmogorov-Smirnov test, and those that achieved normality were analysed using parametric methods. FMPS and FMBS measured before the beginning of each period of experimental mucositis in both groups were compared using the Wilcoxon test. For the other clinical parameters (PI, BoP, PPM, RCAL and PD), ANOVA two way/Tukey test was used to detect differences between groups and periods. Levels of osteo-immunoinflammatory markers between groups and among follow-ups were compared using the Wilcoxon and Friedman test, respectively. An experimental level of significance was determined at 5%.

ELIGIBILITY:
Inclusion Criteria:

* 30 years old or more
* Patients should be smokers (more than 10 cigarettes/day, for at least 2 years),
* present at least a 2-stage unitary screwed implant-supported single-unit crown in the molar or pre-molar region implant connection should be external hexagonal and the implants should be in function at least 12 months
* width of keratinized tissue > 2mm around implants
* The peri-implant tissue should be healthy [probing depth (PD) <4mm with no bleeding on probing (BoP) and no evidence of radiographic bone loss beyond bone remodeling (AAP 2013).
* Patients should be periodontally healthy and present full mouth plaque scores and bleeding score < 20%.

Exclusion Criteria:

* pregnancy
* lactation
* systemic conditions r that could affect the progression of peri-implant diseases and bone metabolism (e.g., immunologic disorders)
* use of long-term administration of anti-inflammatory and immunosuppressive medications antibiotic therapies in the previous 6 months
* individuals that required bone grafts before or alongside the implant surgery history of previous regenerative procedures in the area treated with implant therapy.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Osteo-immunoinflammatory mediators | 21 days
  Levels of interferon (INF), interleukin (IL)-4, IL-17, IL-1β, IL-10, IL-6, IL-23, tumor necrosis factor (TNF)-α (Human Th17 HTH17MAG-14K, Millipore Corporation, Billerica, MA, USA), osteoprotegerin (OPG), osteocalcin (OC), osteopontin (OPN) (Human Bone HBNMAG-51K, Millipore Corporation, Billerica, MA, USA), matrix metalloproteinase (MMP)-2, MMP-9 (Human MMP Panel 2 HMMP2MAG-55K, Millipore Corporation, Billerica, MA, USA), transforming growth factor (TGF)-β (Multi-species TGFβ TGFBMAG-64K, Millipore Corporation, Billerica, MA, USA) and crosslinked telopeptide of type I collagen (ICTP) (Uscn Life Science Inc. Wuhan, Hubei, PRC) in the peri-implant fluid were determined using commercially available kits.

SECONDARY OUTCOMES:
bleeding index | 21 days
  scored using dichotomous index of mucosal marginal bleeding around implants
plaque index | 21 days
  scored using a dichotomous plaque index along the mucosal margin around implants
Position of the peri-implant margin | 21 days
  distance from the stent to the bottom of the peri-implant pocket
Peri-implant probing depth | 21 days
  calculated by deducting PPM from RCAL
Relative clinical attachment level | 21 days
  which was the distance from the stent to the bottom of the peri-implant pocket;

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry - Paulista University UNIP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No